CLINICAL TRIAL: NCT00895310
Title: Assessing PSA Response in Low Dose Ketoconazole in Hormone Refractory Prostate Cancer Patients Who Have Failed at Least One Prior Systemic Chemotherapy Regimen
Brief Title: Use of Low Dose Ketoconazole in Prostate Cancer That Does Not Respond to Hormone Therapy and Prior Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200916901; UCDCC#218 (Other: University of California Davis)
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
Keywords: PSA; Ketoconazole; Prostate Cancer; Hormone Refractory; Chemotherapy Regimen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ketoconazole; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketoconazole and Hydrocortisone (Experimental): Ketoconazole 200mg PO TID + Hydrocortisone 20mg PO Qam, 10mg PO Qpm
  Interventions: Drug: Ketoconazole; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Ketoconazole — Ketoconazole is taken three times a day by mouth.
  Other Names: Nizoral
Drug: Hydrocortisone — Hydrocortisone is taken by mouth 20 mg every morning and 10 mg every evening.
  Other Names: Cortef

SUMMARY:
The purpose of this study is to test the safety of ketoconazole and how well it works after chemotherapy has been used. Ketoconazole at lower doses has been used for fungal infections however has not yet been approved by the Food and Drug Administration for use in prostate cancer. Ketoconazole has been used for many years at high doses for prostate cancer, and this study will be to look at use of lower dose ketoconazole after someone has received chemotherapy. Ketoconazole works by halting the production of steroids in your body, including testosterone, and is thought to work directly on prostate cancer cells in published lab studies.

DETAILED DESCRIPTION:
The aim of the study is to research the response of low dose ketoconazole in hormone refractory prostate cancer (HRPC) patients who have already undergone chemotherapy as part of their prostate cancer treatment. The hypothesis of the study is that HRPC patients who have been previously treated with chemotherapy will demonstrate objective PSA response rates to low dose ketoconazole, comparable to historical response rates reported in chemotherapy-naïve patients. This is a single arm trial, with all participants given ketoconazole 200mg TID, along with hydrocortisone given at 20mg in the morning, 10mg at night daily. Each cycle will consist of 28 days. The subject's study participation will continue until subject experiences disease progression, unacceptable toxicities, withdraws consent from the study or dies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven prostate cancer with a Gleason score available or interpretable.
* Patients must have prostate cancer deemed to be hormone refractory, by progression of measurable or evaluable disease or rising PSA.
* Patients must be >18 years old
* Patients must have received at least one prior chemotherapy regimen >3 weeks prior to initiation of study and patients must have recovered from the side effects of the therapy
* Patients must have an ECOG status of 0-3
* Patients must have normal organ and marrow function, determined within 14 days of registration.
* Patients must have been surgically or medically castrated. If the method of castration was LHRH agonists (leuprolide or goserelin), then the patient must be willing to continue the use of LHRH agonists.
* Patients must have a serum total testosterone level <50 ng/dl
* If the patient has been treated with non-steroidal anti-androgens (flutamide, bicalutamide or nilutamide) or other hormonal treatment (megace or steroids), the patient must have stopped these agents at least 28 days prior to enrollment for flutamide, megace or steroids and at least 42 days prior to enrollment for bicalutamide or nilutamide; and the patients must have demonstrated progression of disease since the agents were suspended.

Exclusion Criteria:

* Patients with any condition that impairs the ability to swallow medications orally
* Patients who are unable to give informed consent
* Patients who have received ketoconazole treatment for prostate cancer in the past
* Patients with other active malignancies in the past 3 years except nonmelanoma skin cancer
* Patients may not be receiving any other investigational agents
* Patients with known hypersensitivity to ketoconazole
* Patients may not be taking certain medications, including terbinafine, astemizole, triazolam, statins (except pravastatin and fluvastatin) and acid suppressive agents (antacids, H2 blockers, PPI) while on ketoconazole, and patients on these medications must agree to discontinue these medications and consider alternative therapies.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N Lara Jr., MD, Principal Investigator — University of California, Davis Health System
Locations (1):
- University of California, Davis Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lo EN, Beckett LA, Pan CX, Robles D, Suga JM, Sands JM, Lara PN Jr. Prospective evaluation of low-dose ketoconazole plus hydrocortisone in docetaxel pre-treated castration-resistant prostate cancer patients. Prostate Cancer Prostatic Dis. 2015 Jun;18(2):144-8. doi: 10.1038/pcan.2015.2. Epub 2015 Feb 10. PMID 25667107

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at a single institution.
Groups:
- Ketoconazole: Ketoconazole 200mg PO (by mouth) TID (three times a day) + Hydrocortisone 20mg PO Qam (every morning), 10mg PO Qpm (every evening)
  Ketoconazole: Ketoconazole is taken three times a day by mouth.
Period: Overall Study
Arm/Group | Ketoconazole
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Ketoconazole: Ketoconazole 200mg PO TID + Hydrocortisone 20mg PO Qam, 10mg PO Qpm
  Ketoconazole: Ketoconazole is taken three times a day by mouth.
Arm/Group | Ketoconazole
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 72 [55 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response (>50% Reduction From Baseline)
Description: Percentage of patients who achieved a clinically significant decline in Prostate Specific Antigen (PSA) after initiation of ketoconazole therapy, defined as a >=50% decrease in PSA.
Time Frame: From date of enrollment, every Cycle (4 weeks), until disease progression, unacceptable toxicities, study withdrawal, or death from any cause, whichever came first, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ketoconazole
Number analyzed (Participants) | 29
Participants | 14

2. Secondary Outcome: PSA Response (>30% From Baseline)
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ketoconazole
Number analyzed (Participants) | 29
Participants | 17

3. Secondary Outcome: Progression Free Survival
Description: Response Evaluation Criteria In Solid Tumors (RECIST) radiographic criteria for progression
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ketoconazole
Number analyzed (Participants) | 29
Days | 138 [80 to 260]

4. Secondary Outcome: Duration of Stable Disease
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Ketoconazole
Number analyzed (Participants) | 29
Days | 123 [2 to 728]

ADVERSE EVENTS:
Time Frame: From the start of treatment until 8-12 weeks after removal from study, assessed for up to 2 years.
Arm/Group | Ketoconazole
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 13/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketoconazole (N=30)
Angina (Cardiac disorders) | 1 (1) — Grade 3
Congestive Heart Failure (Cardiac disorders) | 1 (1) — Grade 3
Myocarditis (Cardiac disorders) | 1 (1) — Grade 3
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Grade 3
Weight Gain (General disorders) | 2 (2) — Grade 3
Fatigue (General disorders) | 1 (1) — Grade 3
Transaminitis (Metabolism and nutrition disorders) | 1 (1) — Grade 3
Hypoantremia (General disorders) | 1 (1) — Grade 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — Grade 3
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3
Syncope (Nervous system disorders) | 1 (1) — Grade 3
Mood Alteration (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) — Grade 3
Pain (General disorders) | 2 (2) — Grade 3
Myocardial Infarction (Cardiac disorders) | 1 (1) — Grade 4
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) — Grade 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes